CLINICAL TRIAL: NCT04383093
Title: Prospective Observational Trial of Combination Therapy of Tadalafil 5mg Plus Tamsulosinmg for Men With Lower Urinary Tract Symptoms and Erectile Dysfunction
Brief Title: Tadalafil Plus Tamsulosin for Male LUTS and ED
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Simone Morselli, MD, University of Florence
Other Study IDs: OSS.15.031/2015
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Prostatic Hyperplasia, Benign; Lower Urinary Tract Symptoms; Erectile Dysfunction; Metabolic Syndrome
Keywords: Tadalafil; Tamsulosin; BPH; LUTS; ED; PDE5-I; Alpha-Blockers; METS
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Erectile Dysfunction; Metabolic Syndrome | interventions — Tadalafil; Tamsulosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combination Therapy: Patients initial assessment included age, waist circumference, blood pressure, clinical laboratory parameters, digital rectal examination. LUTS were evaluated with total IPSS, focusing also on storage, voiding IPSS sub-scores, and IPSS QoL, and Overactive Bladder questionnaire (OAB-q), while ED with IIEF-515. Each patient underwent uroﬂowmetry and postvoid residual volume (PVR) was measured with abdominal ultrasound immediately after voiding. All patients reporting any intake of therapies for LUTS or ED underwent a 4 weeks treatment-free washout period.
  All subjects were treated with tadalafil 5 mg/die plus tamsulosin 0.4 mg/die for 12 weeks. The medications were self-administered every day at the same time, before the night rest, without any limitations or variations of sexual activity timing or food intake. Patients were re-evaluated after 12 weeks of treatment with Uroflowmetry and PVR, IPSS, IPSS QoL, OAB-q and IIEF-5
  Interventions: Drug: Tadalafil 5mg

INTERVENTIONS:
Drug: Tadalafil 5mg — Combination therapy of daily tadalafil plus tamsulosin
  Other Names: Tamsulosin 0.4mg

SUMMARY:
Metabolic Syndrome (MetS) is a complex epidemic disorder with an impact on both lower urinary tract symptoms (LUTS) and erectile dysfunction (ED). Combination therapy of daily tadalafil and tamsulosin may provide relief to both diseases.

Aim of the present study is to assess the impact of combination therapy of Tadalafil 5mg plus Tamsulosin 0.4mg on LUTS and ED, according to presence vs. absence of Mets.

DETAILED DESCRIPTION:
75 Consecutive men presenting with ED and LUTS suggestive of bladder prostatic obstruction were enrolled. Patients were divided into two groups according to MetS presence or absence. All subjects were then treated with tadalafil 5 mg/die plus tamsulosin 0.4 mg/die for 12 weeks. Patients were re-evaluated after 12 weeks of treatment with Uroflowmetry and PVR, IPSS, IPSS QoL, OAB-q and IIEF-5 and comparison were made in and between groups.

ELIGIBILITY:
Inclusion Criteria:

* mild to severe ED (International Index of Erectile Function-Erectile Function-5 <22)
* moderate to severe LUTS (International Prostate Symptom Score >7)

Exclusion Criteria:

* hypersensitivity to tadalaﬁl or tamsulosin
* prostatic cancer or suspected with prostate-speciﬁc antigen (PSA) >4 ng/mL
* bladder lithiasis
* previous prostatic surgery
* urinary tract infection
* neurogenic bladder
* ﬁnasteride or dutasteride use within 3 or 6 months respectively
* clinical history of urethral and/or proven bladder neck obstruction

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 75 Consecutive men presenting with ED and LUTS suggestive of bladder prostatic obstruction (BPO) were screened for the trial. Inclusion criteria were age >40 to 80 years, mild to severe ED (International Index of Erectile Function-Erectile Function-5 <22), moderate to severe LUTS (International Prostate Symptom Score >7), while exclusion criteria were hypersensitivity to tadalaﬁl or tamsulosin, prostatic cancer or suspected with prostate-speciﬁc antigen (PSA) >4 ng/mL, bladder lithiasis, previous prostatic surgery, urinary tract infection, neurogenic bladder, ﬁnasteride or dutasteride use within 3 or 6 months, respectively, clinical history of urethral and/or proven bladder neck obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Lower Urinary Tract Symptoms | Changes from Baseline IPSS at 3 months
  Through IPSS
Lower Urinary Tract Symptoms - Storage | Changes from Baseline OAB-q at 3 months
  Through OAB-q
Erectile Dysfunction | Changes from Baseline IIEF-5 at 3 months
  Through IIEF-5
Flowmetry Maximum Flow | Changes from Baseline Maximum Flow at 3 months
  Through Maximum Flow (ml/s)
Flowmetry Post Void Residual | Changes from Baseline Post Void Residual at 3 months
  Through Post Void Residual (ml)

SECONDARY OUTCOMES:
Combination Therapy Adverse Events | 3 months
  Drug related adverse events were collected
Combination Therapy Compliance | 3 months
  Adherence to therapy - did all the patients took the combination therapy daily
Combination Therapy Tolerability | 3 months
  Measured by the study completion rate by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gacci, MD, Principal Investigator — University of Florence; Arcangelo Sebastianelli, MD, Principal Investigator — University of Florence; Sergio Serni, MD, Principal Investigator — University of Florence

IPD SHARING:
Plan to Share IPD: No